CLINICAL TRIAL: NCT04913532
Title: A Phase II Trial of Evaluation of Acute Toxicity in Hypofractionation With Simultaneous Integrated Boost for Early Breast Cancer
Brief Title: Hypofractionation With Simultaneous Integrated Boost for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Wenjie Ni, Capital Medical University, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-q12
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Surgery; Adjuvant Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionation with SIB (Experimental): Hypofractionation with SIB
  Interventions: Radiation: Hypofractionation with simultaneous integrated boost

INTERVENTIONS:
Radiation: Hypofractionation with simultaneous integrated boost — Hypofractionation with simultaneous integrated boost

SUMMARY:
Simultaneous integrated boost radiotherapy has been investigated in some malignant tumors and appears to be safe and feasible. However, Hypofractionation with simultaneous integrated boost has been investigating in breast cancer.

Investigators initiated this phase II prospective trial to analyse acute toxicity of hypofractionation with simultaneous integrated boost in patients with early breast cancer.

DETAILED DESCRIPTION:
Hypofractionated radiotherapy of the breast 15 × 2.70 Gy with simultaneous integrated boost to the tumor bed (total dose within the boost volume 15 × 3.20 Gy)

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed breast cancer operated by breast conserving surgery with clear margins
* Indication to adjuvant radiotherapy including boost radiotherapy
* Clearly identified primary tumor region preferably by radiopaque clips
* Primary wound healing after breast conserving therapy without signs of infection
* Pre- and/or postoperative chemotherapy and endocrine therapy were permitted when indicated
* Written informed consent

Exclusion Criteria:

* Patients operated by mastectomy
* No indication for boost radiation
* Resection margins positive for disease or insufficient identification of the boost volume
* Indication for radiotherapy of the regional lymph nodes
* History of prior breast or thoracic radiotherapy
* Extended postoperative seroma at the beginning of radiotherapy
* Psychiatric disorders or psychological disabilities thought to adversely affect treatment compliance
* Pregnant or lactating patients and woman of child bearing potential, who lacked effective contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Acute Toxicity | 6 months
  Acute skin radiogenic toxicity grade II or higher according to NCI-CTCAE

SECONDARY OUTCOMES:
Feasibility of the radiation plan | 19 days
  Dose constraints Dmean lung < 10 Gy; Dmean heart < 5 Gy, Dmedian contralateral breast < 4Gy
other acute Toxicity | 0-6 months
  All dimensions of NCI-CTCAE/RTOG

OTHER OUTCOMES:
Skin toxicity (Cosmetic results) | 0 to 6 months
  RTOG

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Ni, MD., Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
No.